CLINICAL TRIAL: NCT03545945
Title: Clinical Advantages of Performing Concomitant Office Hysteroscopy and Endometrial Biopsy in Patients With Oligomenorrhea Seeking Infertility Treatment as Compared to Only Endometrial Biopsy: A Prospective Randomized Study
Brief Title: Hysteroscopy in Chronic Anovulation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to enroll patients
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO 00034165
Record Dates: First submitted 2018-05-22; First posted 2018-06-04 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2019-03

CONDITIONS: Chronic Anovulation

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study arm (Experimental): Patients having office diagnostic hysteroscopy and endometrial biopsy
  Interventions: Procedure: Additional office hysteroscopy; Procedure: Endometrial biopsy
- Control arm (Other): Patients having only endometrial biopsy
  Interventions: Procedure: Endometrial biopsy

INTERVENTIONS:
Procedure: Additional office hysteroscopy — Patients in the study arm will undergo diagnostic office hysteroscopy where they look for any underlying polyp, fibroids or uterine anomaly in addition to endometrial biopsy.
  Arms: Study arm
Procedure: Endometrial biopsy — Patients randomized to endometrial biopsy only group will be prepped with betadine solution and local anesthesia in the form of lidocaine gel placed in the external cervical canal and biopsy will be performed using a Pipelle catheter.

SUMMARY:
Patients with chronic anovulation presenting to the IVF clinic for subfertility treatment are at increased risk of endometrial hyperplasia and carcinoma.They are often subjected to endometrial biopsy to rule out any underlying changes such as endometrial hyperplasia or carcinoma before commencing any further treatment. Literature shows that these group of patients have higher possibility of having underlying uterine abnormality (uterine polyp, fibroid, septum, or adhesion) and if we perform only endometrial biopsy, these structural abnormalities will remain undetected. And presence of uterine abnormalities lead to difficulty in implantation, which eventually leads to lower success rate of infertility treatment.

WE propose that performing simultaneous office hysteroscopy followed by endometrial biopsy in such patients will lead to higher detection of uterine structural abnormalities and obtaining endometrial tissue to rule out hyperplasia or carcinoma. The concern for clinicians at times is that performing both the procedures together will lead to higher pain perception during the procedure. But with the introduction of flexible hysteroscope which has a diameter of 3.5 mm we hypothesize that the pain of performing office hysteroscopy with endometrial biopsy and performing endometrial biopsy alone will be equivalent. Meanwhile, hysteroscopy will lead lead to detection of underlying uterine pathology and help us in taking directed biopsies.

DETAILED DESCRIPTION:
Patients with subfertility due to hormonal disorders are at increased risk of endometrial cancer and hyperplasia . Such conditions are associated with chronic anovulation, obesity and/or hyperinsulinemia. Presumably, the mechanism relates to constant, unrelenting estrogen stimulation of the endometrium, predisposing to abnormal patterns of growth. Hence, patients with long standing anovulation presenting for infertility evaluation, are often subjected to endometrial biopsy to rule out any underlying hyperplasia or malignancy.

The polycystic ovary syndrome (PCOS) is the most obvious and common condition associated with chronic anovulation. It is characterized by hyperandrogenism, ovulatory dysfunction, and polycystic ovarian morphologic features. Based on National Institutes of Health (i.e. hyperandrogenism plus ovulatory dysfunction), "classic" polycystic ovary syndrome affects 10% of women of reproductive age but the prevalence may be twice under the broader Rotterdam criteria . Women with PCOS are at increased risk of infertility, endometrial hyperplasia and cancer. The risk of endometrial cancer in a woman with PCOS is reported to be 2.7 times higher than someone without this syndrome. Other uncommon conditions associated with chronic anovulation are Cushing's syndrome, congenital adrenal hyperplasia secondary to 21 hydroxylase deficiency, thyroid or liver disorder leading to decreased clearance of estrogen from the body. Similarly, obese postmenopausal women are also at increased risk for developing endometrial cancer.

In these patients, elevated plasma levels of androgen precursors increase estrogen level through aromatization of androgens in adipose tissue. In addition, it has been seen that non cycling patients with grossly increased endometrial thickness (greater than 12 mm) are also at high risk of endometrial hyperplasia. So these are the indications, which warrants patients to undergo endometrial biopsy. Literature shows that the prevalence of minor intrauterine abnormalities identified at hysteroscopy in cases with a normal transvaginal sonography (TVS) can be as high as 20-40%. Similarly, the prevalence of unsuspected uterine cavity abnormalities, diagnosed in an unselected group of patients undergoing IVF can be 11%. In this study, they identified endometrial polyps in 6% women, submucous myomas in 1%, intrauterine adhesions (2%), and septa (2%) . Another study also reports 16% intracavitary lesion in patients with infertility. It has been seen that in an IVF population, obesity (BMI >30) is also an independent risk factor for developing endometrial polyps. The prevalence of polyps in patients with BMI > 30 is 52% as compared to 15% among patients with BMI <30. Similarly, PCOS patients also show a higher incidence of endometrial polyp (29%) diagnosed by hysteroscopy as compared to the nonPCOS population and the presence of 2 or more such polyps is associated with significant premalignant or malignant condition. So, missing the diagnosis of polyps in PCOS patients renders them to higher risk of developing malignancy in future. With this background, an important clinical question is if it is clinically justified to combine office hysteroscopy and endometrial biopsy as part of the comprehensive evaluation of these patients? It is possible that prompt diagnosis and treatment of these unsuspected uterine abnormalities could optimize the condition of the uterine environment and thereby the outcome of treatment.

In spite of all the advantages office hysteroscopy offers, one of the reasons for avoiding office hysteroscopy has been the apprehension that adding office hysteroscopy will lead to higher pain score. But based on our literature review we propose that adding flexible office hysteroscopy to endometrial biopsy will not lead to any increase in pain score. In routine practice, endometrial biopsy is usually performed with "Pipelle" and is a simple office procedure. It is an excellent tool for evaluating the histopathology of the endometrium. The mean pain score during endometrial biopsy is 3 in a VAS scale of 1-10 with only 6.7% patients reporting severe pain . In a more recent study, the pain score during endometrial biopsy has been reported to be 6.2, which is higher than the previous reports. Similarly, office hysteroscopy is also a simple procedure with high patient acceptability and safety. The pain score reported during office hysteroscopy using flexible scope range from 2.3 -3. During traditional hysteroscopy where speculum and tenaculum is used, the pain score has been reported to be as high as 5.3. In fact, a comparative study of endometrial biopsy and office hysteroscopy showed that the pain score is higher during endometrial biopsy (5.1) as compared to diagnostic hysteroscopy (2.7). Hence, it seems very reasonable to add office hysteroscopy to endometrial biopsy for patients undergoing endometrial evaluation. This combined approach will have better diagnostic yield without increasing the pain perception.

ELIGIBILITY:
Inclusion Criteria:

All consecutive reproductive age female patients (aged 15-45) presenting to IVF clinic for medically indicated endometrial biopsy for evaluation of endometrial pathology with ability to provide written informed consent.

Sub-fertile women presenting with history of chronic anovulation and in addition meets any one of the criteria mentioned below:

1. Women with ≤ 3 menstrual cycle per year.
2. Women with oligomenorrhea and BMI >30.
3. Women with oligomenorrhea and endometrial thickness >12 mm measured during transvaginal sonography -

Exclusion Criteria:

1. Patients unable to provide informed consent.
2. Patients presenting to USF-IVF clinic for evaluation of infertility but endometrial biopsy is not deemed clinically relevant based on assessment by provider.
3. Patients refusing participation in lieu of additional procedure.
4. Patients are already known to have existing uterine abnormality diagnosed by ultrasound. -

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Detection of unsuspected underlying uterine abnormalities. (i.e. polyp, fibroids, septum and/or adhesion) | 1 year
  The primary outcome of the study is to determine whether performing office hysteroscopy in addition to endometrial biopsy in subfertile patients who are at risk of endometrial hyperplasia or cancer, enhances the chances of detection of unsuspected underlying uterine abnormalities. (i.e. polyp, fibroids, septum and/or adhesion).

SECONDARY OUTCOMES:
Pain score (evaluated on VAS scale) | 1 year
  Our secondary outcome is to compare the pain score (evaluated on VAS scale) between patients who are having office hysteroscopy in addition to endometrial biopsy with patients who are having endometrial biopsy alone (VAS scale).

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Florida, Department of Obstetrics and Gynecology, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klip H, Burger CW, Kenemans P, van Leeuwen FE. Cancer risk associated with subfertility and ovulation induction: a review. Cancer Causes Control. 2000 Apr;11(4):319-44. doi: 10.1023/a:1008921211309. PMID 10843444
- [Background] Legro RS. Diagnostic criteria in polycystic ovary syndrome. Semin Reprod Med. 2003 Aug;21(3):267-75. doi: 10.1055/s-2003-43304. PMID 14593549